CLINICAL TRIAL: NCT00672139
Title: Open-Label Extension Study To Assess The Safety Of A Fixed Dose Of Subcutaneous Methylnaltrexone In Subjects With Advanced Illness And Opioid-Induced Constipation
Brief Title: Safety of Subcutaneous Methylnaltrexone for Opioid-Induced Constipation in Patients With Advanced Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3200K1-4001; B2541006
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Opioid-Induced Constipation
Keywords: Opioid-Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylnaltrexone bromide (Experimental): Methylnaltrexone subcutaneously as needed no more than 1 dose in a 24-hour period for a maximum of 10 weeks in this study.
  Subjects received 0.6 mL (12 mg) every other day if weight ≥ 62kg; or 0.4 mL (8 mg) every other day if weight between 38 and <62 kg. Subjects with impaired kidney function received reduced doses according to instructions in the Relistor prescribing information.
  Interventions: Drug: Methylnaltrexone bromide

INTERVENTIONS:
Drug: Methylnaltrexone bromide
  Other Names: Relistor

SUMMARY:
This is an open-label, multicenter extension of study 3200K1-4000-WW that will evaluate the safety of methylnaltrexone. This drug will be administered by subcutaneous injection and will be tested in late stage, advanced illness patients who have constipation caused by opioid pain relievers. This study will last 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Has completed study 3200K1-4000-WW, including 2 weeks of therapy and completion of all post baseline efficacy, safety, and health outcomes assessments.
* Is receiving opioids on a regular schedule, not just as needed to control pain.
* Likely to continue to need treatment of OIC for the duration of participation in the study.

Exclusion Criteria:

* Has a suspected mechanical gastrointestinal obstruction, fecal impaction, or clinically important active diverticular disease as determined by the investigator.
* Currently using an opioid antagonist or partial antagonist.
* Has any other clinically important abnormalities such that risk to patient of participation outweighs the potential benefit of therapy as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-07; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Bortey, Study Director — Bausch Health Americas, Inc.
Locations (41):
- United States (23):
  - Salix Investigational Site, Mobile, Alabama
  - Salix Investigational Site, Laguna Hills, California
  - Salix Investigational Site, Lancaster, California
  - Salix Investigational Site, Aurora, Colorado
  - Salix Investigational Site, Auburndale, Florida
  - Salix Investigational Site, Hudson, Florida
  - Salix Investigational Site, Lakeland, Florida
  - Salix Investigational Site, Miami Springs, Florida
  - Salix Investigational Site, Ruskin, Florida
  - Salix Investigational Site, Sebring, Florida
  - Salix Investigational Site, Tampa, Florida
  - Salix Investigational Site, Temple Terrace, Florida
  - Salix Investigational Site, Orange, New Jersey
  - Salix Investigational Site, Flat Rock, North Carolina
  - Salix Investigational Site, Winston-Salem, North Carolina
  - Salix Investigational Site, Cleveland, Ohio
  - Salix Investigational Site, Philadelphia, Pennsylvania
  - Salix Investigational Site, Austin, Texas
  - Salix Investigational Site, Houston, Texas
  - Salix Investigational Site, American Fork, Utah
  - Salix Investigational Site, Orem, Utah
  - Salix Investigational Site, Provo, Utah
  - Salix Investigational Site, Madison, Wisconsin
- Australia (3):
  - Salix Investigational Site, Coburg, Victoria
  - Salix Investigational Site, East Melbourne, Victoria
  - Salix Investigational Site, Adelaide
- Salix Investigational Site, Leuven, Belgium
- Canada (5):
  - Salix Investigational Site, Edmonton, Alberta
  - Salix Investigational Site, Hamilton, Ontario
  - Salix Investigational Site, London, Ontario
  - Salix Investigational Site, Montreal, Quebec
  - Salix Investigational Site, Québec, Quebec
- Salix Investigational Site, Montpellier, France
- Salix Investigational Site, Berlin, Germany
- Italy (3):
  - Salix Investigational Site, L’Aquila
  - Salix Investigational Site, Milan
  - Salix Investigational Site, Roma
- Pfizer Investigational Site, Mexico City DF, Mexico
- Portugal (2):
  - Salix Investigational Site, Almada
  - Salix Investigational Site, Porto
- Salix Investigational Site, Cheltenham, Gloucestershire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients participated in this study at sites in Australia, Belgium, Brazil, Canada, France, Germany, Italy, Mexico, Spain, Sweden, the United Kingdom, and the United States.
Pre-assignment Details: The main eligibility criteria for this study were completion of 2 weeks of therapy and all post-baseline efficacy, safety, and health outcomes assessments in lead-in study MNTX4000 and an anticipated continued need for treatment of opioid-induced constipation.
Groups:
- Methylnaltrexone Bromide 8 mg: Methylnaltrexone subcutaneously as needed no more than 1 dose in a 24-hour period for a maximum of 10 weeks in this study.
  Subjects received 0.4 mL (8 mg) every other day if weight between 38 and <62 kg. Subjects with impaired kidney function received reduced doses according to instructions in the Relistor prescribing information.
- Methylnaltrexone Bromide 12 mg: Methylnaltrexone subcutaneously as needed no more than 1 dose in a 24-hour period for a maximum of 10 weeks in this study.
  Subjects received 0.6 mL (12 mg) every other day if weight ≥ 62kg. Subjects with impaired kidney function received reduced doses according to instructions in the Relistor prescribing information.
Period: Overall Study
Arm/Group | Methylnaltrexone Bromide 8 mg | Methylnaltrexone Bromide 12 mg
Started | 57 (Three of 60 enrolled subjects did not receive study drug.) | 92 (Four of 96 enrolled subjects did not receive study drug.)
Completed | 27 | 47
Not Completed | 30 | 45
Not completed — Death | 14 | 23
Not completed — Withdrawal by Subject | 2 | 11
Not completed — Adverse Event | 4 | 7
Not completed — Physician Decision | 2 | 0
Not completed — Lack of Efficacy | 4 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — hospice discharge, caregiver requests | 3 | 2

BASELINE CHARACTERISTICS:
Population: The analysis population included subjects who received study drug and had laxation data and drug administration data. Two subjects in the 12 mg/day group had no drug administration data and were not included in efficacy analyses (but they were included in baseline characteristics and safety analyses).
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylnaltrexone Bromide 8 mg | Methylnaltrexone Bromide 12 mg | Total
Number analyzed (Participants) | 57 | 92 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 46 | 70
  >=65 years | 33 | 46 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.07 (14.29) | 64.59 (11.98) | 65.92 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 33 | 77
  Male | 13 | 59 | 72
Underlying Advanced Illness [Number; unit: Participants]
  Cancer | 36 | 49 | 85
  Pulmonary disease | 7 | 18 | 25
  Cardiovascular disease | 4 | 15 | 19
  Neurologic disease | 3 | 3 | 6
  Other | 7 | 7 | 14
Weight [Number; unit: participants]
  38 to < 62 kg | 54 | 0 | 54
  ≥ 62 kg | 3 | 92 | 95
Glomerular filtration rate [Number; unit: participants]
  < 30 mL/min/1.73 m^2 | 2 | 0 | 2
  ≥ 30 mL/min/1.73 m^2 | 54 | 89 | 143
  Missing | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Laxations Per Subject Within 24 Hours of Dosing Per Week.
Description: This was defined as the total number of days with a laxation (ie, a bowel movement) within 24 hours after dosing in each 7-day interval after the start of dosing. Results shown are the ranges (lowest and highest weekly values) of mean (± standard deviation) numbers of laxations within 24 hours of dosing per week during the 10-week treatment period for each group.
Time Frame: 10 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Number of laxations
Arm/Group | Methylnaltrexone Bromide 8 mg | Methylnaltrexone Bromide 12 mg
Number analyzed (Participants) | 57 | 90
Number of laxations
  Lowest weekly average # laxations/week | 1.7 (1.5) | 2.4 (2.3)
  Highest weekly average # laxations/week | 2.6 (2.4) | 3.4 (3.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 10-week treatment period.
Description: Adverse events were collected by non-systematic (patient reports) and systematic methods (investigator examinations and lab tests). For both adverse events tables, a subject reporting more than one adverse event for a particular MedDRA preferred term or system organ class was counted only once for that MedDRA preferred term or system organ class.
Arm/Group | Methylnaltrexone Bromide 8 mg | Methylnaltrexone Bromide 12 mg
Serious Adverse Events (participants affected / at risk) | 22/57 | 37/92
Other Adverse Events (participants affected / at risk) | 45/57 | 60/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone Bromide 8 mg (N=57) | Methylnaltrexone Bromide 12 mg (N=92)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Disease progression (General disorders) | 15 | 22
General physical health deterioration (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone Bromide 8 mg (N=57) | Methylnaltrexone Bromide 12 mg (N=92)
Abdominal pain (Gastrointestinal disorders) | 13 | 21
Diarrhea (Gastrointestinal disorders) | 11 | 12
Dysphagia (Gastrointestinal disorders) | 3 | 3
Flatulence (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 5 | 14
Vomiting (Gastrointestinal disorders) | 4 | 5
Asthenia (General disorders) | 10 | 8
Chest pain (General disorders) | 1 | 5
Disease progression (General disorders) | 4 | 4
Fatigue (General disorders) | 3 | 3
Oedema peripheral (General disorders) | 10 | 13
Pyrexia (General disorders) | 1 | 10
Urinary tract infection (Infections and infestations) | 6 | 7
Contusion (Injury, poisoning and procedural complications) | 7 | 1
Fall (Injury, poisoning and procedural complications) | 8 | 12
Laceration (Injury, poisoning and procedural complications) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 5
Dizziness (Nervous system disorders) | 4 | 6
Lethargy (Nervous system disorders) | 4 | 3
Agitation (Psychiatric disorders) | 5 | 7
Anxiety (Psychiatric disorders) | 4 | 7
Confusional state (Psychiatric disorders) | 9 | 11
Restlessness (Psychiatric disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Rales (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less